CLINICAL TRIAL: NCT02689206
Title: A 29-day, Randomized, Double-blinded, Placebo-controlled, Parallel-group, Multi-center Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Three-times Weekly Dosing of GSK1278863 in Hemodialysis-dependent Subjects With Anemia Associated With Chronic Kidney Disease Who Are Switched From a Stable Dose of an Erythropoiesis-stimulating Agent
Brief Title: Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Three-times Weekly Dosing of GSK1278863 in Hemodialysis-dependent Subjects With Anemia Associated With Chronic Kidney Disease Who Are Switched From a Stable Dose of an Erythropoiesis-stimulating Agent
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204836; 2015-004790-32 (EudraCT Number)
Record Dates: First submitted 2016-02-11; First posted 2016-02-23 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Anaemia
Keywords: Chronic kidney disease; Efficacy; Erythropoiesis-stimulating agent; GSK1278863; Safety; Hemodialysis-dependent anemia; Pharmacokinetics
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- GSK1278863 10 mg (Experimental): Subject will receive 10 mg of GSK1278863 three-times weekly for 4 weeks (up to 29 days).
  Interventions: Drug: GSK1278863
- GSK1278863 15 mg (Experimental): Subject will receive 15 mg of GSK1278863 three-times weekly for 4 weeks (up to 29 days).
  Interventions: Drug: GSK1278863
- GSK1278863 25 mg (Experimental): Subject will receive 25 mg of GSK1278863 three-times weekly for 4 weeks (up to 29 days).
  Interventions: Drug: GSK1278863
- GSK1278863 30 mg (Experimental): Subject will receive 30 mg of GSK1278863 three-times weekly for 4 weeks (up to 29 days).
  Interventions: Drug: GSK1278863
- Placebo (Placebo Comparator): Subject will receive GSK1278863 matching placebo three-times weekly for 4 weeks (up to 29 days).
  Interventions: Drug: GSK1278863 matching Placebo

INTERVENTIONS:
Drug: GSK1278863 — GSK1278863 will be supplied as a round, biconvex, 10 millimeter (mm) white film coated tablet with the unit dose strength of 5 mg and 25 mg.
  Arms: GSK1278863 10 mg; GSK1278863 15 mg; GSK1278863 25 mg; GSK1278863 30 mg
Drug: GSK1278863 matching Placebo — GSK1278863 matching placebo will be supplied as a round, biconvex, 10 mm white film coated tablet.
  Arms: Placebo

SUMMARY:
GSK1278863 is an orally available, hypoxia-inducible factor - prolyl hydroxylase inhibitor, currently being investigated as a treatment for anemia associated with chronic kidney disease. GSK1278863 has been given as a once daily regimen in clinical studies to date. However, physicians in countries that use a three-times weekly hemodialysis schedule prefer to give the anemia medicine at the same time as the dialysis session. This study will test how well GSK1278863 can maintain hemoglobin levels when given three-times weekly, for 29 days.

This study will describe the relationship between hemoglobin and GSK1278863 given three-times weekly. The data from this study will allow for conversion of once daily doses to three-times weekly doses.

ELIGIBILITY:
Inclusion Criteria:

* More than or equal to 18 years of age, at the time of signing the informed consent.
* Hemoglobin: Stable Hemoglobin 9.0 - 11.5 gram per deciliter (g/dL).
* Dialysis frequency: On hemodialysis (HD, hemofiltration or hemodiafiltration) three to five times weekly for at least 4 weeks prior to Day -28 Screening through Day 29.
* Dialysis adequacy: A single pool Kt/Vurea of >=1.2 based on a historical value obtained within the prior three months in order to ensure the adequacy of dialysis. If Kt/Vurea is not available, then an average of the last 2 values of urea reduction ratio (URR) of at least 65 percent. NOTE: Only needs confirming at Day -28.
* Erythropoiesis-stimulating agent (ESA)dose: Treated with the same ESA (epoetins or their biosimilars, or darbepoetin or methoxy polyethylene glycol [PEG]-epoetin beta) with total weekly dose varying by no more than 50 percent during the 4 weeks prior to Day -28.
* Iron replacement therapy: Subjects may be on stable maintenance oral or intravenous (IV) (<=100 milligram (mg)/week) iron supplementation. If subjects are on oral or IV iron, then doses must be stable for the 4 weeks prior to Day -28, during the screening phase, and through the 29 days of treatment.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in study protocol.

Exclusion Criteria:

* Dialysis modality: Planned change from HD to peritoneal dialysis within the study time period.
* Renal transplant: Planned for living-related kidney transplant.
* High ESA dose: An epoetin dose of >=360 international unit (IU)/kilogram (kg)/week IV or >=250 IU/kg/week subcutaneous (SC) or darbepoetin dose of >=1.8 microgram (mcg)/kg/week IV or SC or methoxy PEG-epoetin beta dose of >= 2.2 mcg/kg/week within the prior 8 weeks through Day 1 (randomization).
* Administration of methoxy PEG-epoetin beta within the prior 4 weeks through Day 1 (randomization).
* Myocardial infarction or acute coronary syndrome: Within the 8 weeks prior to Screening through Day 1 (randomization).
* Stroke or transient ischemic attack: Within 8 weeks prior to Screening though Day 1 (randomization).
* Heart failure: Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system diagnosed prior to Screening through Day 1 (randomization).
* Correction of Q-T Interval using Bazett's formula (QTcB): QTcB >500 millisecond (msec) or QTcB >530 msec in subjects with Bundle Branch Block. There is no correction of Q-T Interval (QTc) exclusion for subjects with a predominantly paced rhythm.
* Inflammatory disease: Active chronic inflammatory disease that could impact erythropoiesis (e.g., scleroderma, systemic lupus erythematosis, rheumatoid arthritis, celiac disease) diagnosed prior to Screening through Day 1 (randomization).
* Hematological disease: Any hematological disease including those affecting platelets, white or red blood cells (e.g., sickle cell anemia, myelodysplastic syndromes, hematological malignancy, myeloma, hemolytic anemia and thalassemia), coagulation disorders (e.g., antiphospholipid syndrome, Protein C or S deficiency), or any other cause of anemia of chronic disease other than renal disease diagnosed prior to Screening though Day 1 (randomization).
* Liver disease: Current liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or evidence at Screening of abnormal liver function tests [alanine transaminase (ALT) or aspartate transaminase (AST) >2x upper limit of normal (ULN) or total bilirubin >1.5xULN]; or other hepatic abnormalities that in the opinion of the investigator would preclude the subject from participating in the study.

NOTE: Those with Hepatitis B or Hepatitis C are eligible provided these exclusions are not met.

* Major surgery: Major surgery (excluding vascular access surgery) within the 8 weeks prior to Screening, during the Screening phase, or planned during the study.
* Transfusion: Blood transfusion within the 8 weeks prior to Screening, during the Screening phase or an anticipated need for blood transfusion during the study.
* Gastrointestinal (GI) Bleeding: Evidence of actively bleeding peptic, duodenal, or esophageal ulcer disease OR clinically significant GI bleeding within the 8 weeks prior to Screening through Day 1 (randomization).
* Acute Infection: Clinical evidence of acute infection or history of infection requiring IV antibiotic therapy within the 4 weeks prior to Screening through Day 1 (randomization). NOTE: IV antibiotics as prophylaxis are allowed.
* Malignancy: History of malignancy within the two years prior to randomization or currently receiving treatment for cancer, or has a known >=4 centimeter complex kidney cyst (i.e. Bosniak Category II F, III of IV). NOTE: ONLY exception is squamous cell or basal cell carcinoma of the skin that has been definitively treated >=8 weeks prior to Screening.
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product
* Drugs and supplements: Use of any prescription or non-prescription drugs or dietary supplements that are prohibited (as per protocol) from Screening until the Follow-up Visit.
* Prior investigational product exposure: The Subject has participated in a clinical trial and has received an experimental investigational product within the prior 30 days from Screening through Day 1 (randomization).
* Other conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the subject at unacceptable risk, which may affect study compliance or prevent understanding of the aims or investigational procedures or possible consequences of the study.
* Females ONLY: A female subject is not eligible to participate if she is pregnant [as confirmed by a positive serum human chorionic gonadotrophin (hCG) test for females of reproductive potential (FRP) only], breastfeeding, and if of reproductive potential does not agree to follow one of the options listed in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP.
* Vitamin B12: At or below the lower limit of the reference range (may rescreen in a minimum of 8 weeks).
* Folate: <2.0 nanogram (ng) per millilitre (mL) (4.5 nanomole/liter [L]) (may rescreen in a minimum of 4 weeks).
* Ferritin: <100 ng/mL (<100 mcg/L).
* Transferrin saturation (TSAT): <20 percent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2017-01-25 (Actual); Study Completion 2017-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- United States (7):
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, San Dimas, California
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Greenbelt, Maryland
  - GSK Investigational Site, Roseville, Michigan
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, The Bronx, New York
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
- Germany (4):
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Darmstadt
- Russia (7):
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Mytischi
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Yaroslavl
- Spain (13):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Granollers, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Lleida
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Manises (Valencia)
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, San Sebastián de los Reyes
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valladolid

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20174

REFERENCES:
- [Background] Bailey CK, Caltabiano S, Cobitz AR, Huang C, Mahar KM, Patel VV. A randomized, 29-day, dose-ranging, efficacy and safety study of daprodustat, administered three times weekly in patients with anemia on hemodialysis. BMC Nephrol. 2019 Oct 16;20(1):372. doi: 10.1186/s12882-019-1547-z. PMID 31619187
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants on Hemodialysis (HD) with anemia associated with chronic kidney disease (CKD) switching from Erythropoiesis-Stimulating Agent (ESA) treatment were recruited in this randomized, dose-ranging study. Participants with hemoglobin (Hgb) values between 9.0- 11.5 grams per deciliter (g/dL) were considered as eligible for recruitment.
Pre-assignment Details: A total of 211 participants were screened; of which 108 were screen failures and 103 were randomized to receive at least one dose of either placebo or 10, 15, 25 or 30 milligrams (mg) of daprodustat (dapro). One participant who was randomized to the placebo group, erroneously received 25 mg dapro treatment throughout the 29-day treatment period
Groups:
- Placebo: Randomized participants received placebo tablet via oral route three times weekly for 29 days.
- Dapro 10 mg: Randomized participants received dapro 10 mg tablet via oral route three times weekly for 29 days.
- Dapro 15 mg: Randomized participants received dapro 15 mg tablet via oral route three times weekly for 29 days.
- Dapro 25 mg: Randomized participants received dapro 25 mg tablet via oral route three times weekly for 29 days.
- Dapro 30 mg: Randomized participants received dapro 30 mg tablet via oral route three times weekly for 29 days
Period: Overall Study
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Started | 20 | 20 | 20 | 21 | 22
Completed | 17 | 19 | 16 | 17 | 14
Not Completed | 3 | 1 | 4 | 4 | 8
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 1 | 2
Not completed — Other: Reached stopping criteria | 0 | 1 | 2 | 3 | 4
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg | Total
Number analyzed (Participants) | 20 | 20 | 20 | 21 | 22 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (13.06) | 63.6 (16.98) | 59.5 (12.26) | 67.2 (15.22) | 65.4 (13.97) | 63.4 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 6 | 9 | 8 | 42
  Male | 9 | 12 | 14 | 12 | 14 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race customized: African American/African Heritage | 6 | 6 | 7 | 5 | 6 | 30
  Race customized: American Indian Or Alaskan Native | 0 | 1 | 0 | 0 | 1 | 2
  Race customized: Asian - Central/South Asian Heritage | 0 | 1 | 1 | 0 | 0 | 2
  Race customized: Native Hawaiian Or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Race customized: White- Arabic/North African Heritage | 0 | 0 | 0 | 1 | 0 | 1
  Race customized: White-White/Caucasian/European Heritage | 14 | 12 | 12 | 14 | 15 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hgb Levels at Day 29
Description: Blood samples were collected from participants for measurement of Hgb values. Baseline is the average of Hgb measured at Week -2 and Day 1 visits. Change from Baseline at Day 29 was defined as post dose value at Day 29 minus Baseline value. The analysis was performed on intent-to-treat (ITT) Population which comprised of all randomized participants who received at least one dose of study treatment, had a Baseline and at least one corresponding on treatment assessment, including Hgb.
Time Frame: Baseline and Day 29
Population: ITT Population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 17 | 19 | 16 | 17 | 15
g/dL | -0.61 (0.646) | -0.19 (1.750) | -0.13 (1.088) | 0.64 (1.453) | 0.55 (1.167)
Statistical Analysis 1: Comparison: Placebo vs Dapro 10 mg; Test type: Other; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.31 to 1.45] — Analysis using a Repeated Measures Model with terms included for baseline, treatment, time and treatment*time. Model-adjusted treatment difference of dapro 10 mg arm from Placebo along with 95 percent CI are presented
Statistical Analysis 2: Comparison: Placebo vs Dapro 15 mg; Test type: Other; Mean Difference (Final Values) = 0.51, 95% CI 2-sided [-0.40 to 1.42] — Analysis using a Repeated Measures Model with terms included for baseline, treatment, time and treatment*time. Model-adjusted treatment difference of dapro 15 mg arm from Placebo along with 95 percent CI are presented
Statistical Analysis 3: Comparison: Placebo vs Dapro 25 mg; Test type: Other; Mean Difference (Final Values) = 1.47, 95% CI 2-sided [0.59 to 2.35] — Analysis using a Repeated Measures Model with terms included for baseline, treatment, time and treatment*time. Model-adjusted treatment difference of dapro 25 mg arm from Placebo along with 95 percent CI are presented
Statistical Analysis 4: Comparison: Placebo vs Dapro 30 mg; Test type: Other; Mean Difference (Final Values) = 1.67, 95% CI 2-sided [0.77 to 2.57] — Analysis using a Repeated Measures Model with terms included for baseline, treatment, time and treatment*time. Model-adjusted treatment difference of dapro 30 mg arm from Placebo along with 95 percent CI are presented

2. Secondary Outcome: Maximum Observed Change From Baseline in Plasma Erythropoietin (EPO)
Description: Blood samples were collected at Day 1, Day 15 and Day 29 for pharmacodynamic analysis of effect of dapro three times weekly dose regimens on EPO. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. The change from Baseline at each given post-Baseline time point was calculated and the maximum change from Baseline was determined.
Time Frame: Baseline and up to Day 29
Population: ITT Population
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 18 | 20 | 18 | 21 | 20
International unit per liter (IU/L) | 53.761 (132.6875) | 2.255 (84.8921) | 73.369 (95.9772) | 302.529 (469.8312) | 477.644 (388.9757)

3. Secondary Outcome: Maximum Observed Percent Change From Baseline in Vascular Endothelial Growth Factor (VEGF)
Description: Blood samples were collected at Day 1, Day 15 and Day 29 for pharmacodynamic analysis of effect of dapro three times weekly dose regimens on VEGF. Day 1 values were considered as Baseline values. The percent change from Baseline at each given post-Baseline time point was calculated (expressed as geometric mean) and the maximum percent change from Baseline was determined.
Time Frame: Baseline and up to Day 29
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per liter (ng/L)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 18 | 20 | 18 | 21 | 20
Nanograms per liter (ng/L) | 20.35 [-0.48 to 45.55] | 43.75 [16.44 to 77.45] | 32.16 [-4.77 to 83.41] | 53.34 [17.17 to 100.68] | 76.09 [34.89 to 129.88]

4. Secondary Outcome: Percent Change From Baseline in Hepcidin at Day 29
Description: Blood samples were collected at Day 1, Day 15 and Day 29 for pharmacodynamic analysis of effect of dapro three times weekly dose regimens on hepcidin. Day 1 values were considered as Baseline values. The Percent change from Baseline at Day 29 post-Baseline time point was calculated and expressed as geometric mean and the maximum change from Baseline was determined.
Time Frame: Baseline and Day 29
Population: ITT Population
Measure: Geometric Mean (95% Confidence Interval); unit: Micrograms per liter (µg/L)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 17 | 19 | 15 | 17 | 15
Micrograms per liter (µg/L) | 27.81 [-12.68 to 87.08] | 35.37 [-1.13 to 85.34] | 3.83 [-17.85 to 31.24] | -36.74 [-49.91 to -20.12] | -36.09 [-57.24 to -4.48]

5. Secondary Outcome: Change From Baseline in Hematocrit Levels
Description: Blood samples were collected at Day 1, Day 15 and Day 29 for pharmacodynamic analysis of effect Dapro three times weekly dose regimens on hematocrit. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-dose visit values minus Baseline value. The change from Baseline at Day 29 post-Baseline time point was calculated.
Time Frame: Baseline and Day 29
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 16 | 19 | 14 | 16 | 15
Proportion of red blood cells in blood | -0.0218 (0.02469) | -0.0127 (0.05396) | -0.0149 (0.05379) | 0.0150 (0.04511) | 0.0215 (0.03852)

6. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count
Description: Blood samples were collected at Day 1, Day 15 and Day 29 for pharmacodynamic analysis of effect Dapro three times weekly dose regimens on RBC count. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-dose visit values minus Baseline value. The change from Baseline at Day 29 post-Baseline time point was calculated.
Time Frame: Baseline and Day 29
Population: ITT Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 16 | 19 | 14 | 16 | 15
10^12 cells/L | -0.19 (0.263) | -0.12 (0.494) | -0.13 (0.500) | 0.12 (0.420) | 0.15 (0.342)

7. Secondary Outcome: Change From Baseline in Reticulocyte Count
Description: Blood samples were collected at Day 1, Day 15 and Day 29 for pharmacodynamic analysis of effect Dapro three times weekly dose regimens on reticulocyte count. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. The change from Baseline at Day 29 post-Baseline time point was calculated.
Time Frame: Baseline and Day 29
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Percentage of reticulocyte
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 16 | 18 | 14 | 16 | 15
Percentage of reticulocyte | -0.08 (0.848) | -0.11 (0.803) | -0.04 (0.581) | 0.43 (0.547) | 0.09 (0.695)

8. Secondary Outcome: Change From Baseline in Reticulocyte Hemoglobin (CHr)
Description: Blood samples were collected at Day 1, Day 15 and Day 29 for pharmacodynamic analysis of effect Dapro three times weekly dose regimens on CHr. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. The change from Baseline at Day 29 post-Baseline time point was calculated.
Time Frame: Baseline and Day 29
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Picograms (pg)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 16 | 19 | 14 | 16 | 15
Picograms (pg) | -0.15 (1.375) | 0.23 (1.335) | 0.26 (1.103) | 0.23 (1.040) | 0.59 (1.436)

9. Secondary Outcome: Area Under the Curve (AUC) From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-t]) and AUC From Time Zero to Infinity (AUC[0-inf]) of Dapro
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of dapro. The data from each PK sampling day was combined to generate a single profile, and normalized to a 24-hour period to create a "Day 1" profile for non-compartmental analysis (NCA). Metabolite plasma concentrations were analyzed but PK parameters could not be calculated as the metabolites were partially eliminated through dialysis and the dialysis start and end times were not consistent on both PK days. Therefore, a representative metabolite PK profile could not be generated. The analysis was performed on PK Population, which comprised of all participants from whom a PK sample has been obtained and analyzed. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Pre-dose on Day 1; 6-10 hours, 7-11 hours, 8-12 hours, 9-13 hours post dose on Day 15; pre-dose and 1, 2, 3 hours post-dose on Day 29
Population: PK Population. One participant who was randomized to the placebo group, erroneously received 25mg daprodustat treatment throughout the 29-day treatment period. This subject is counted within the daprodustat 25mg treatment group for all PK population and safety population analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour into nanograms/milliliter (h*ng/mL)
Arm/Group | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 20 | 20 | 22 | 22
hour into nanograms/milliliter (h*ng/mL)
  AUC (0-t); n= 19, 15, 16, 14: number analyzed (Participants) | 19 | 15 | 16 | 14
  AUC (0-t); n= 19, 15, 16, 14 | 311.7 (91.4) | 416.7 (168.6) | 513.9 (396.1) | 1010 (92.3)
  AUC (0-inf); n= 12, 9, 8, 11: number analyzed (Participants) | 12 | 9 | 8 | 11
  AUC (0-inf); n= 12, 9, 8, 11 | 348.2 (78.2) | 383.5 (142.7) | 1214 (41.6) | 1369 (59.3)

10. Secondary Outcome: Maximum Observed Concentration of Dapro in Plasma (Cmax)
Description: Blood samples were collected at indicated time points for PK analysis of dapro. The data from each PK sampling day was combined to generate a single profile, and normalized to a 24-hour period to create a "Day 1" profile for NCA. Metabolite plasma concentrations were analyzed but PK parameters could not be calculated as the metabolites were partially eliminated through dialysis and the dialysis start and end times were not consistent on both PK days. Therefore, a representative metabolite PK profile could not be generated.
Time Frame: as for outcome 9
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 15 | 16 | 14
ng/mL | 140.0 (104.0) | 141.4 (248.8) | 246.9 (311.5) | 387.3 (99.4)

11. Secondary Outcome: Time to Reach Cmax (Tmax) and Apparent Terminal Half-life (t1/2) of Dapro
Description: Blood samples were collected at indicated time points for PK analysis of dapro. The data from each PK sampling day was combined to generate a single profile, and normalized to a 24-hour period to create a "Day 1" profile for NCA. Metabolite plasma concentrations were analyzed but PK parameters could not be calculated as the metabolites were partially eliminated through dialysis and the dialysis start and end times were not consistent on both PK days. Therefore, a representative metabolite PK profile could not be generated. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour
Arm/Group | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 20 | 20 | 22 | 22
Hour
  Tmax; n= 19, 15, 16, 14: number analyzed (Participants) | 19 | 15 | 16 | 14
  Tmax; n= 19, 15, 16, 14 | 2.456 (78.9) | 2.106 (82.1) | 2.297 (96.5) | 1.718 (58.0)
  T1/2; n= 12, 9, 8, 11: number analyzed (Participants) | 12 | 9 | 8 | 11
  T1/2; n= 12, 9, 8, 11 | 2.086 (50.0) | 1.886 (62.3) | 1.418 (58.4) | 2.897 (38.7)

12. Secondary Outcome: Number of Participants Who Discontinued Study Treatment
Description: Reasons of study treatment discontinuation included adverse events (AEs), protocol deviation, participants reached protocol defined stopping criteria, physician decision and withdrawal by participants. Number of participants who discontinued study treatment are presented. Analysis was performed on Safety Population which comprised of all participants who received at least one dose of study treatment.
Time Frame: Up to Day 43
Population: Safety Population. One participant who was randomized to the placebo group, erroneously received 25mg daprodustat treatment throughout the 29-day treatment period. This subject is counted within the daprodustat 25mg treatment group for all PK population and safety population analyses.
Measure: Number; unit: Participants
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Participants
  AEs | 0 | 0 | 1 | 0 | 1
  Protocol deviation | 1 | 0 | 0 | 1 | 2
  Participant reached stopping criteria | 0 | 1 | 2 | 3 | 4
  Physician decision | 1 | 0 | 0 | 0 | 0
  Withdrawal by subject | 1 | 0 | 1 | 0 | 0

13. Secondary Outcome: Number of Participants With AEs and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability, is a congenital anomaly/ birth effect, other situations and is associated with liver injury or impaired liver function.
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Participants
  Any AE | 10 | 10 | 6 | 7 | 7
  Any SAE | 4 | 3 | 2 | 1 | 3

14. Secondary Outcome: Sodium, Potassium, Glucose, Calcium, Phosphate Levels in Blood at Indicated Time Points
Description: Serum sodium, potassium, glucose, corrected calcium and phosphate levels were assessed as a clinical chemistry laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Millimoles per liter (mmol/L)
  Sodium; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Sodium; Day 1; n= 18, 20, 20, 22, 22 | 138.8 (2.85) | 138.1 (2.31) | 138.7 (2.83) | 139.4 (2.38) | 138.4 (1.76)
  Sodium; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Sodium; Day 15; n= 17, 20, 18, 22, 20 | 137.7 (3.16) | 137.5 (2.72) | 138.1 (1.60) | 138.0 (2.36) | 137.2 (1.74)
  Sodium; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Sodium; Day 29; n= 17, 19, 18, 19, 17 | 137.8 (3.96) | 136.8 (2.70) | 137.9 (2.85) | 138.8 (2.74) | 137.1 (2.46)
  Sodium; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Sodium; Day 43; n= 15, 20, 18, 21, 21 | 139.2 (2.88) | 138.1 (1.77) | 137.9 (2.37) | 138.8 (2.02) | 137.6 (1.88)
  Potassium; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Potassium; Day 1; n= 18, 20, 20, 22, 22 | 4.68 (0.840) | 4.73 (0.768) | 4.64 (0.826) | 4.79 (0.514) | 4.83 (0.685)
  Potassium; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Potassium; Day 15; n= 17, 20, 18, 22, 20 | 4.72 (0.763) | 4.77 (0.542) | 4.57 (0.635) | 4.82 (0.765) | 4.80 (0.791)
  Potassium; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Potassium; Day 29; n= 17, 19, 18, 19, 17 | 4.78 (0.919) | 4.87 (0.751) | 4.57 (0.472) | 4.86 (0.619) | 4.96 (0.941)
  Potassium; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Potassium; Day 43; n= 15, 20, 18, 21, 21 | 4.69 (0.951) | 4.68 (0.562) | 4.59 (0.657) | 4.76 (0.752) | 4.80 (0.946)
  Glucose; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Glucose; Day 1; n= 18, 20, 20, 22, 22 | 6.66 (3.088) | 6.66 (2.716) | 6.41 (3.507) | 7.05 (2.491) | 8.95 (5.012)
  Glucose; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Glucose; Day 15; n= 17, 20, 18, 22, 20 | 7.89 (3.425) | 7.16 (2.844) | 7.03 (3.236) | 7.26 (2.852) | 8.67 (4.198)
  Glucose; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Glucose; Day 29; n= 17, 19, 18, 19, 17 | 8.21 (4.951) | 7.49 (3.949) | 7.21 (3.953) | 7.77 (4.621) | 8.75 (5.708)
  Glucose; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Glucose; Day 43; n= 15, 20, 18, 21, 21 | 6.93 (3.126) | 6.72 (2.965) | 7.09 (3.533) | 6.27 (1.958) | 8.93 (4.280)
  Calcium corrected; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Calcium corrected; Day 1; n= 18, 20, 20, 22, 22 | 2.286 (0.2116) | 2.270 (0.1244) | 2.241 (0.1675) | 2.219 (0.1589) | 2.215 (0.1163)
  Calcium corrected; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Calcium corrected; Day 15; n= 17, 20, 18, 22, 20 | 2.261 (0.1698) | 2.219 (0.1252) | 2.213 (0.1723) | 2.188 (0.1360) | 2.203 (0.1111)
  Calcium corrected; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Calcium corrected; Day 29; n= 17, 19, 18, 19, 17 | 2.205 (0.1431) | 2.248 (0.1352) | 2.244 (0.1577) | 2.198 (0.1343) | 2.225 (0.1810)
  Calcium corrected; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Calcium corrected; Day 43; n= 15, 20, 18, 21, 21 | 2.251 (0.1582) | 2.235 (0.1593) | 2.271 (0.1823) | 2.201 (0.1206) | 2.256 (0.1473)
  Phosphate; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Phosphate; Day 1; n= 18, 20, 20, 22, 22 | 1.608 (0.5143) | 1.528 (0.5557) | 1.498 (0.5265) | 1.318 (0.3647) | 1.566 (0.4269)
  Phosphate; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Phosphate; Day 15; n= 17, 20, 18, 22, 20 | 1.621 (0.4221) | 1.710 (0.3912) | 1.642 (0.5021) | 1.348 (0.3138) | 1.645 (0.4785)
  Phosphate; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Phosphate; Day 29; n= 17, 19, 18, 19, 17 | 1.709 (0.5872) | 1.592 (0.4121) | 1.644 (0.5322) | 1.453 (0.4489) | 1.550 (0.3575)
  Phosphate; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Phosphate; Day 43; n= 15, 20, 18, 21, 21 | 1.550 (0.5828) | 1.460 (0.4550) | 1.472 (0.4240) | 1.412 (0.4441) | 1.398 (0.4718)

15. Secondary Outcome: Albumin and Protein Levels in Blood at Indicated Tme Points
Description: Serum albumin and protein levels were assessed as a clinical chemistry laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
grams per liter (g/L)
  Albumin; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Albumin; Day 1; n= 18, 20, 20, 22, 22 | 37.6 (2.89) | 38.6 (2.46) | 38.7 (3.84) | 38.8 (2.22) | 38.1 (3.52)
  Albumin; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Albumin; Day 15; n= 17, 20, 18, 22, 20 | 38.1 (2.68) | 38.1 (2.65) | 38.4 (3.42) | 38.4 (2.52) | 37.2 (3.01)
  Albumin; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Albumin; Day 29; n= 17, 19, 18, 19, 17 | 36.5 (3.22) | 37.2 (3.26) | 37.6 (3.62) | 37.4 (2.17) | 36.9 (4.15)
  Albumin; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Albumin; Day 43; n= 15, 20, 18, 21, 21 | 37.1 (2.85) | 38.1 (3.02) | 37.9 (3.95) | 39.0 (3.11) | 37.5 (2.86)
  Protein; Day 1; n= 18, 20 ,20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Protein; Day 1; n= 18, 20 ,20, 22, 22 | 67.3 (4.90) | 66.9 (5.42) | 67.4 (4.89) | 66.4 (5.16) | 65.7 (4.65)
  Protein; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Protein; Day 15; n= 17, 20, 18, 22, 20 | 68.1 (4.87) | 66.5 (4.88) | 67.3 (4.28) | 65.6 (5.13) | 64.3 (4.70)
  Protein; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Protein; Day 29; n= 17, 19, 18, 19, 17 | 66.1 (4.52) | 65.7 (4.75) | 66.0 (4.51) | 65.5 (6.50) | 65.3 (5.30)
  Protein; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Protein; Day 43; n= 15, 20, 18, 21, 21 | 67.2 (4.25) | 67.4 (5.14) | 66.8 (4.02) | 66.7 (7.70) | 66.6 (6.34)

16. Secondary Outcome: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Alkaline Phosphatase (Alk. Phosph) Levels in Blood at Indicated Time Points
Description: Serum ALT, AST and alk. phosph. levels were assessed as a clinical chemistry laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: Safety Population One participant who was randomized to the placebo group, erroneously received 25mg daprodustat treatment throughout the 29-day treatment period. This subject is counted within the daprodustat 25mg treatment group for all PK population and safety population analyses.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
IU/L
  ALT; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  ALT; Day 1; n= 18, 20, 20, 22, 22 | 12.6 (9.36) | 13.4 (7.51) | 14.6 (11.39) | 10.7 (5.75) | 11.5 (5.94)
  ALT; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  ALT; Day 15; n= 17, 20, 18, 22, 20 | 16.5 (13.80) | 13.9 (10.58) | 12.4 (7.87) | 11.9 (6.58) | 8.4 (2.11)
  ALT; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  ALT; Day 29; n= 17, 19, 18, 19, 17 | 24.4 (32.34) | 12.8 (6.43) | 12.2 (6.40) | 10.9 (5.67) | 8.6 (3.12)
  ALT; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  ALT; Day 43; n= 15, 20, 18, 21, 21 | 14.3 (8.55) | 13.8 (8.03) | 12.8 (6.89) | 13.1 (5.19) | 11.2 (5.57)
  AST; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  AST; Day 1; n= 18, 20, 20, 22, 22 | 14.9 (5.58) | 14.2 (5.19) | 17.2 (12.31) | 14.4 (5.85) | 13.6 (3.63)
  AST; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  AST; Day 15; n= 17, 20, 18, 22, 20 | 17.1 (7.30) | 14.3 (5.67) | 15.0 (7.72) | 15.4 (6.33) | 12.4 (2.89)
  AST; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  AST; Day 29; n= 17, 19, 18, 19, 17 | 26.8 (30.04) | 13.8 (5.01) | 16.0 (8.44) | 15.0 (6.35) | 13.5 (3.12)
  AST; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  AST; Day 43; n= 15, 20, 18, 21, 21 | 15.9 (6.65) | 14.9 (6.07) | 17.2 (11.40) | 15.7 (6.31) | 14.3 (4.76)
  Alk. phosph; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Alk. phosph; Day 1; n= 18, 20, 20, 22, 22 | 97.0 (33.07) | 112.3 (74.61) | 106.8 (84.85) | 99.4 (47.26) | 115.4 (72.35)
  Alk. phosph; Day 15; n= 17, 20, 18, 22,20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Alk. phosph; Day 15; n= 17, 20, 18, 22,20 | 102.4 (34.70) | 115.4 (73.37) | 114.5 (82.29) | 101.5 (56.44) | 110.0 (62.65)
  Alk. phosph.; Day 29; n= 17, 19, 18, 19,17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Alk. phosph.; Day 29; n= 17, 19, 18, 19,17 | 94.1 (35.07) | 120.2 (81.15) | 109.2 (83.14) | 93.5 (42.92) | 120.4 (67.51)
  Alk. phosph.; Day 43; n= 15, 20, 18, 21,21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Alk. phosph.; Day 43; n= 15, 20, 18, 21,21 | 96.5 (34.12) | 117.6 (76.61) | 113.8 (78.69) | 116.2 (96.02) | 108.6 (50.49)

17. Secondary Outcome: Bilirubin, Direct Bilirubin and Indirect Bilirubin Levels in Blood at Indicated Time Points
Description: Serum bilirubin, direct bilirubin and indirect bilirubin levels were assessed as a clinical chemistry laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Micromoles per liter (µmol/L)
  Bilirubin; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Bilirubin; Day 1; n= 18, 20, 20, 22, 22 | 6.6 (1.65) | 7.8 (3.11) | 6.6 (1.31) | 6.5 (1.10) | 7.2 (2.44)
  Bilirubin; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Bilirubin; Day 15; n= 17, 20, 18, 22, 20 | 6.7 (3.08) | 7.1 (2.29) | 7.2 (2.67) | 6.5 (1.10) | 7.8 (2.24)
  Bilirubin; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Bilirubin; Day 29; n= 17, 19, 18, 19, 17 | 6.8 (2.24) | 6.9 (1.93) | 7.6 (2.12) | 6.5 (1.47) | 7.8 (2.44)
  Bilirubin; Day 43; n= 15, 20 ,18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Bilirubin; Day 43; n= 15, 20 ,18, 21, 21 | 6.0 (1.07) | 7.0 (2.38) | 7.2 (2.07) | 6.5 (1.25) | 7.5 (2.44)
  Direct bilirubin; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Direct bilirubin; Day 1; n= 18, 20, 20, 22, 22 | 1.8 (1.17) | 1.9 (0.79) | 2.0 (1.12) | 1.9 (0.75) | 2.4 (1.33)
  Direct bilirubin; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Direct bilirubin; Day 15; n= 17, 20, 18, 22, 20 | 1.5 (1.66) | 2.2 (0.62) | 2.4 (1.29) | 1.8 (0.85) | 2.6 (1.14)
  Direct bilirubin; Day 29; n= 17, 19, 18, 19,17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Direct bilirubin; Day 29; n= 17, 19, 18, 19,17 | 2.5 (2.29) | 1.6 (1.07) | 2.7 (0.97) | 1.8 (0.63) | 2.4 (1.46)
  Direct bilirubin; Day 43; n= 15, 20, 18, 21,21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Direct bilirubin; Day 43; n= 15, 20, 18, 21,21 | 1.3 (1.23) | 1.9 (0.45) | 2.3 (0.77) | 1.7 (0.72) | 2.3 (1.31)
  Indirect bilirubin; Day 1; n= 18, 20, 20, 22, 22: number analyzed (Participants) | 18 | 20 | 20 | 22 | 22
  Indirect bilirubin; Day 1; n= 18, 20, 20, 22, 22 | 4.8 (1.22) | 5.9 (2.94) | 4.6 (0.94) | 4.6 (1.14) | 4.8 (1.92)
  Indirect bilirubin; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Indirect bilirubin; Day 15; n= 17, 20, 18, 22, 20 | 5.2 (2.01) | 4.9 (2.10) | 4.8 (1.83) | 4.7 (0.98) | 5.2 (1.77)
  Indirect bilirubin; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Indirect bilirubin; Day 29; n= 17, 19, 18, 19, 17 | 4.4 (2.03) | 5.4 (1.64) | 4.9 (1.57) | 4.7 (1.52) | 5.4 (1.70)
  Indirect bilirubin; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Indirect bilirubin; Day 43; n= 15, 20, 18, 21, 21 | 4.7 (0.98) | 5.1 (2.38) | 4.9 (1.41) | 4.8 (1.48) | 5.2 (1.73)

18. Secondary Outcome: Change From Baseline in Sodium, Potassium, Glucose, Calcium and Phosphate Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including sodium, potassium, glucose, calcium and phosphate. Change from Baseline in clinical chemistry parameters at Day 15, Day 29 and Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Mmol/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Mmol/L
  Sodium; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Sodium; Day 15; n= 17, 20, 18, 22, 20 | -0.9 (2.73) | -0.6 (2.62) | -0.5 (2.64) | -1.4 (2.06) | -1.0 (2.13)
  Sodium; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Sodium; Day 29; n= 17, 19, 18, 19, 17 | -1.1 (2.26) | -1.2 (3.08) | -0.9 (2.26) | -0.5 (2.82) | -1.2 (2.70)
  Sodium; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Sodium; Day 43; n= 15, 20, 18, 21, 21 | 0.7 (2.06) | 0.1 (2.35) | -0.6 (2.28) | -0.5 (2.60) | -0.6 (2.23)
  Potassium; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Potassium; Day 15; n= 17, 20, 18, 22, 20 | 0.04 (0.462) | 0.05 (0.526) | -0.09 (1.099) | 0.03 (0.944) | -0.08 (0.635)
  Potassium; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Potassium; Day 29; n= 17, 19, 18, 19, 17 | 0.20 (0.744) | 0.05 (0.660) | -0.14 (0.651) | 0.02 (0.640) | 0.11 (0.673)
  Potassium; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Potassium; Day 43; n= 15, 20, 18, 21, 21 | 0.04 (0.565) | -0.05 (0.674) | -0.06 (1.004) | -0.06 (0.579) | -0.02 (0.932)
  Glucose; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Glucose; Day 15; n= 17, 20, 18, 22, 20 | 1.14 (3.339) | 0.51 (2.959) | 0.45 (1.740) | 0.21 (1.620) | -0.03 (2.364)
  Glucose; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Glucose; Day 29; n= 17, 19, 18, 19, 17 | 1.48 (3.771) | 0.70 (3.756) | 0.73 (1.135) | 0.61 (4.188) | -0.36 (3.786)
  Glucose; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Glucose; Day 43; n= 15, 20, 18, 21, 21 | 0.23 (1.335) | 0.06 (3.072) | 0.52 (1.383) | -0.81 (2.516) | -0.12 (3.619)
  Calcium; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Calcium; Day 15; n= 17, 20, 18, 22, 20 | -0.011 (0.1227) | -0.051 (0.1354) | -0.026 (0.1439) | -0.031 (0.0956) | -0.010 (0.0912)
  Calcium; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Calcium; Day 29; n= 17, 19, 18, 19, 17 | -0.054 (0.1486) | -0.025 (0.1129) | -0.009 (0.1556) | -0.012 (0.0939) | 0.001 (0.1019)
  Calcium; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Calcium; Day 43; n= 15, 20, 18, 21, 21 | -0.015 (0.1576) | -0.035 (0.1261) | 0.018 (0.1852) | 0.001 (0.0742) | 0.033 (0.1489)
  Phosphate; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Phosphate; Day 15; n= 17, 20, 18, 22, 20 | -0.091 (0.4051) | 0.183 (0.5184) | 0.111 (0.5715) | 0.030 (0.3268) | 0.095 (0.3367)
  Phosphate; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Phosphate; Day 29; n= 17, 19, 18, 19, 17 | 0.091 (0.3882) | 0.011 (0.4932) | 0.069 (0.4950) | 0.129 (0.2740) | -0.026 (0.3653)
  Phosphate; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Phosphate; Day 43; n= 15, 20, 18, 21, 21 | -0.067 (0.4337) | -0.068 (0.5324) | -0.053 (0.5400) | 0.102 (0.3433) | -0.117 (0.5117)

19. Secondary Outcome: Change From Baseline in Albumin and Protein Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including albumin and protein. Change from Baseline in clinical chemistry parameters at Day 15, Day 29 and Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
g/L
  Albumin; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Albumin; Day 15; n= 17, 20, 18, 22, 20 | 0.8 (1.60) | -0.5 (1.64) | 0.2 (2.24) | -0.5 (1.44) | -1.0 (2.34)
  Albumin; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Albumin; Day 29; n= 17, 19, 18, 19, 17 | -0.5 (2.24) | -1.3 (2.03) | -0.7 (2.00) | -1.3 (1.85) | -0.9 (1.76)
  Albumin; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Albumin; Day 43; n= 15, 20, 18, 21, 21 | 0.1 (2.00) | -0.6 (2.14) | -0.7 (2.22) | 0.1 (3.85) | -0.3 (1.74)
  Protein; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Protein; Day 15; n= 17, 20, 18, 22, 20 | 0.8 (2.97) | -0.4 (3.25) | 0.3 (3.65) | -0.7 (2.35) | -1.5 (3.03)
  Protein; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Protein; Day 29; n= 17, 19, 18, 19, 17 | -1.1 (4.26) | -0.8 (3.82) | -1.2 (2.90) | -1.0 (3.28) | 0.1 (2.56)
  Protein; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Protein; Day 43; n= 15, 20, 18, 21, 21 | -0.1 (4.19) | 0.6 (4.38) | -0.9 (3.17) | 0.3 (4.84) | 1.2 (3.95)

20. Secondary Outcome: Change From Baseline in ALT, AST, Alk. Phosph. Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including ALT, AST, Alk. phosph. Change from Baseline in clinical chemistry parameters at Day 15, Day 29 and Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
IU/L
  ALT; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  ALT; Day 15; n= 17, 20, 18, 22, 20 | 3.6 (9.59) | 0.5 (5.65) | -3.1 (5.53) | 1.1 (4.79) | -3.4 (5.52)
  ALT; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  ALT; Day 29; n= 17, 19, 18, 19, 17 | 11.8 (32.39) | -0.9 (4.65) | -3.4 (9.83) | -0.2 (3.87) | -3.6 (4.72)
  ALT; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  ALT; Day 43; n= 15, 20, 18, 21, 21 | 0.9 (4.32) | 0.4 (5.29) | -2.5 (8.97) | 2.2 (4.08) | -0.4 (3.69)
  AST; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  AST; Day 15; n= 17, 20, 18, 22, 20 | 2.3 (5.70) | 0.1 (2.45) | -2.7 (6.29) | 1.0 (5.26) | -1.6 (3.32)
  AST; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  AST; Day 29; n= 17, 19, 18, 19, 17 | 11.5 (30.64) | -0.3 (3.30) | -1.8 (5.60) | 0.9 (3.60) | -0.3 (3.67)
  AST; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  AST; Day 43; n= 15, 20, 18, 21, 21 | 0.6 (3.94) | 0.7 (2.49) | -0.6 (7.99) | 1.5 (3.71) | 0.7 (3.41)
  Alk.phosph.; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Alk.phosph.; Day 15; n= 17, 20, 18, 22, 20 | 3.2 (10.28) | 3.2 (16.13) | 2.7 (29.73) | 2.1 (17.23) | -4.7 (18.90)
  Alk.phosph.; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Alk.phosph.; Day 29; n= 17, 19, 18, 19, 17 | -0.4 (19.31) | 5.1 (19.09) | -0.9 (30.13) | 0.9 (13.47) | -1.2 (28.60)
  Alk.phosph.; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Alk.phosph.; Day 43; n= 15, 20, 18, 21, 21 | -1.5 (17.01) | 5.4 (21.34) | 2.7 (31.96) | 18.0 (66.44) | -8.4 (56.06)

21. Secondary Outcome: Change From Baseline in Bilirubin, Direct Bilirubin, Indirect Bilirubin Levels
Description: Blood samples were collected from participants to evaluate clinical chemistry parameters including bilirubin, direct bilirubin and indirect bilirubin. Change from Baseline in clinical chemistry parameters at Day 15, Day 29 and Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
µmol/L
  Bilirubin; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Bilirubin; Day 15; n= 17, 20, 18, 22, 20 | 0.2 (1.56) | -0.7 (1.49) | 0.8 (2.07) | 0.0 (1.38) | 0.5 (1.93)
  Bilirubin; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Bilirubin; Day 29; n= 17, 19, 18, 19, 17 | 0.2 (0.97) | -0.3 (1.20) | 1.0 (1.41) | 0.1 (1.56) | 0.2 (0.97)
  Bilirubin; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Bilirubin; Day 43; n= 15, 20, 18, 21, 21 | -0.1 (0.52) | -0.8 (1.51) | 0.6 (2.04) | 0.1 (1.34) | 0.4 (1.36)
  Direct bilirubin; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Direct bilirubin; Day 15; n= 17, 20, 18, 22, 20 | -0.1 (1.11) | 0.3 (0.73) | 0.6 (0.92) | -0.1 (0.97) | 0.2 (1.11)
  Direct bilirubin; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Direct bilirubin; Day 29; n= 17, 19, 18, 19, 17 | 0.7 (1.86) | -0.3 (1.00) | 0.7 (0.97) | -0.1 (1.05) | -0.1 (1.50)
  Direct bilirubin; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Direct bilirubin; Day 43; n= 15, 20, 18, 21, 21 | -0.1 (1.19) | 0.0 (0.92) | 0.3 (1.03) | -0.2 (1.08) | -0.1 (1.34)
  Indirect bilirubin; Day 15; n= 17, 20, 18, 22, 20: number analyzed (Participants) | 17 | 20 | 18 | 22 | 20
  Indirect bilirubin; Day 15; n= 17, 20, 18, 22, 20 | 0.4 (1.46) | -1.0 (1.38) | 0.2 (1.80) | 0.1 (1.44) | 0.3 (1.75)
  Indirect bilirubin; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Indirect bilirubin; Day 29; n= 17, 19, 18, 19, 17 | -0.5 (1.66) | 0.0 (1.15) | 0.3 (1.71) | 0.2 (1.62) | 0.4 (1.46)
  Indirect bilirubin; Day 43; n= 15, 20, 18, 21, 21: number analyzed (Participants) | 15 | 20 | 18 | 21 | 21
  Indirect bilirubin; Day 43; n= 15, 20, 18, 21, 21 | 0.0 (1.07) | -0.8 (1.64) | 0.2 (1.66) | 0.3 (1.82) | 0.5 (1.40)

22. Secondary Outcome: Leukocytes, Neutrophils, Basophils, Eosinophils,Lymphocytes, Monocytes, Platelet Levels in Blood at Indicated Time Points
Description: Serum leukocytes, neutrophils, basophils, eosinophils, lymphocytes, monocytes and platelet levels were assessed as a clinical hematology laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
10^12 cells/L
  Leukocytes; Day 1; n= 18, 19, 19, 20, 21: number analyzed (Participants) | 18 | 19 | 19 | 20 | 21
  Leukocytes; Day 1; n= 18, 19, 19, 20, 21 | 6.28 (1.750) | 6.07 (1.601) | 5.88 (1.510) | 6.44 (1.595) | 5.90 (1.825)
  Leukocytes; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Leukocytes; Day 15; n= 17, 19, 17, 21, 21 | 7.01 (2.140) | 5.85 (1.720) | 6.21 (1.918) | 6.52 (1.427) | 5.87 (1.961)
  Leukocytes; Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Leukocytes; Day 29; n= 16, 19, 17, 18, 17 | 6.66 (1.707) | 6.59 (1.890) | 5.88 (1.685) | 6.33 (1.820) | 6.11 (2.574)
  Leukocytes; Day 43; n= 16, 20, 19, 20, 19: number analyzed (Participants) | 16 | 20 | 19 | 20 | 19
  Leukocytes; Day 43; n= 16, 20, 19, 20, 19 | 7.05 (2.006) | 7.25 (2.520) | 6.00 (1.694) | 6.77 (2.547) | 6.42 (2.010)
  Neutrophils; Day 1; n= 18, 19, 19, 20, 21: number analyzed (Participants) | 18 | 19 | 19 | 20 | 21
  Neutrophils; Day 1; n= 18, 19, 19, 20, 21 | 4.030 (1.6128) | 4.097 (1.5763) | 3.522 (1.3492) | 3.954 (1.4097) | 3.785 (1.5024)
  Neutrophils; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Neutrophils; Day 15; n= 17, 19, 17, 21, 21 | 4.666 (1.8113) | 3.887 (1.5659) | 3.707 (1.6592) | 4.346 (1.2240) | 4.129 (1.6604)
  Neutrophils; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Neutrophils; Day 29; n= 16, 18, 17, 17, 15 | 4.123 (1.2229) | 4.591 (1.9586) | 3.522 (1.4546) | 3.978 (1.7026) | 4.224 (2.2017)
  Neutrophils; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Neutrophils; Day 43; n= 16, 20, 19, 19, 19 | 4.687 (1.8919) | 5.049 (2.3848) | 3.545 (1.4027) | 4.477 (2.2480) | 4.343 (1.6235)
  Basophils; Day 1; n= 18, 19, 19, 20, 21: number analyzed (Participants) | 18 | 19 | 19 | 20 | 21
  Basophils; Day 1; n= 18, 19, 19, 20, 21 | 0.018 (0.0131) | 0.016 (0.0134) | 0.025 (0.0174) | 0.028 (0.0204) | 0.017 (0.0142)
  Basophils; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Basophils; Day 15; n= 17, 19, 17, 21, 21 | 0.027 (0.0214) | 0.026 (0.0161) | 0.022 (0.0139) | 0.025 (0.0325) | 0.024 (0.0140)
  Basophils; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Basophils; Day 29; n= 16, 18, 17, 17, 15 | 0.035 (0.0462) | 0.021 (0.0128) | 0.021 (0.0150) | 0.024 (0.0111) | 0.027 (0.0315)
  Basophils; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Basophils; Day 43; n= 16, 20, 19, 19, 19 | 0.028 (0.0217) | 0.018 (0.0136) | 0.020 (0.0183) | 0.025 (0.0204) | 0.024 (0.0130)
  Eosinophils; Day 1; n= 18, 19, 19, 20, 21: number analyzed (Participants) | 18 | 19 | 19 | 20 | 21
  Eosinophils; Day 1; n= 18, 19, 19, 20, 21 | 0.189 (0.1946) | 0.174 (0.1593) | 0.184 (0.1696) | 0.196 (0.2310) | 0.240 (0.2115)
  Eosinophils; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Eosinophils; Day 15; n= 17, 19, 17, 21, 21 | 0.161 (0.1245) | 0.166 (0.1804) | 0.192 (0.2355) | 0.187 (0.2186) | 0.186 (0.1914)
  Eosinophils; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Eosinophils; Day 29; n= 16, 18, 17, 17, 15 | 0.176 (0.1917) | 0.149 (0.0950) | 0.145 (0.1136) | 0.237 (0.2785) | 0.185 (0.0798)
  Eosinophils; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Eosinophils; Day 43; n= 16, 20, 19, 19, 19 | 0.216 (0.2458) | 0.210 (0.1969) | 0.232 (0.2727) | 0.243 (0.2670) | 0.217 (0.1899)
  Lymphocytes; Day 1; n= 18, 19, 19, 20, 21: number analyzed (Participants) | 18 | 19 | 19 | 20 | 21
  Lymphocytes; Day 1; n= 18, 19, 19, 20, 21 | 1.631 (0.4264) | 1.393 (0.4587) | 1.739 (0.6964) | 1.747 (0.7325) | 1.442 (0.4998)
  Lymphocytes; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Lymphocytes; Day 15; n= 17, 19, 17, 21, 21 | 1.735 (0.6699) | 1.416 (0.5670) | 1.842 (0.7381) | 1.526 (0.6697) | 1.206 (0.4609)
  Lymphocytes; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Lymphocytes; Day 29; n= 16, 18, 17, 17, 15 | 1.870 (0.7427) | 1.427 (0.4187) | 1.775 (0.6767) | 1.612 (0.5775) | 1.181 (0.3418)
  Lymphocytes; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Lymphocytes; Day 43; n= 16, 20, 19, 19, 19 | 1.648 (0.5294) | 1.509 (0.4386) | 1.736 (0.3916) | 1.721 (0.6644) | 1.399 (0.5562)
  Monocytes; Day 1; n= 18, 19, 20, 20, 21: number analyzed (Participants) | 18 | 19 | 20 | 20 | 21
  Monocytes; Day 1; n= 18, 19, 20, 20, 21 | 0.401 (0.1511) | 0.396 (0.1591) | 0.435 (0.2703) | 0.518 (0.2077) | 0.421 (0.1722)
  Monocytes; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Monocytes; Day 15; n= 17, 19, 17, 21, 21 | 0.420 (0.2243) | 0.352 (0.1457) | 0.436 (0.2402) | 0.446 (0.2085) | 0.384 (0.2160)
  Monocytes; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Monocytes; Day 29; n= 16, 18, 17, 17, 15 | 0.444 (0.2076) | 0.457 (0.1503) | 0.403 (0.1385) | 0.600 (0.3465) | 0.426 (0.2628)
  Monocytes; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Monocytes; Day 43; n= 16, 20, 19, 19, 19 | 0.461 (0.1878) | 0.459 (0.1916) | 0.461 (0.2614) | 0.513 (0.2739) | 0.429 (0.2047)
  Platelet; Day 1; n= 16, 19, 20, 19, 21: number analyzed (Participants) | 16 | 19 | 20 | 19 | 21
  Platelet; Day 1; n= 16, 19, 20, 19, 21 | 219.0 (65.04) | 189.9 (36.70) | 198.0 (71.03) | 196.0 (61.12) | 192.3 (70.85)
  Platelet; Day 15; n= 17, 18, 17, 20, 21: number analyzed (Participants) | 17 | 18 | 17 | 20 | 21
  Platelet; Day 15; n= 17, 18, 17, 20, 21 | 205.4 (63.00) | 175.4 (44.08) | 198.5 (73.65) | 194.8 (49.08) | 181.5 (66.59)
  Platelet; Day 29; n= 16, 19, 17, 17, 17: number analyzed (Participants) | 16 | 19 | 17 | 17 | 17
  Platelet; Day 29; n= 16, 19, 17, 17, 17 | 198.1 (76.39) | 174.7 (52.50) | 187.5 (62.66) | 198.9 (55.07) | 194.8 (81.57)
  Platelet; Day 43; n= 15, 20, 19, 21, 20: number analyzed (Participants) | 15 | 20 | 19 | 21 | 20
  Platelet; Day 43; n= 15, 20, 19, 21, 20 | 220.8 (61.57) | 195.8 (68.33) | 188.6 (69.28) | 194.1 (50.35) | 170.0 (44.61)

23. Secondary Outcome: Mean Corpuscular Hemoglobin (MCH) Levels in Blood at Indicated Time Points
Description: Serum MCH levels were assessed as a clinical hematology laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Pg
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Pg
  Day 1; n= 18, 19, 20, 20, 21: number analyzed (Participants) | 18 | 19 | 20 | 20 | 21
  Day 1; n= 18, 19, 20, 20, 21 | 31.19 (2.538) | 30.95 (1.889) | 30.19 (2.145) | 30.70 (1.781) | 31.46 (1.942)
  Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Day 15; n= 17, 19, 17, 21, 21 | 30.83 (2.100) | 2.100 (1.866) | 30.74 (1.476) | 30.85 (1.619) | 31.70 (2.315)
  Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Day 29; n= 16, 19, 17, 18, 17 | 30.97 (2.290) | 31.60 (2.194) | 30.56 (2.236) | 31.16 (1.729) | 31.68 (2.224)
  Day 43; n= 16, 20, 19, 21, 20: number analyzed (Participants) | 16 | 20 | 19 | 21 | 20
  Day 43; n= 16, 20, 19, 21, 20 | 30.86 (1.992) | 31.04 (1.870) | 30.49 (2.155) | 30.67 (1.846) | 31.84 (2.143)

24. Secondary Outcome: Mean Corpuscular Hemoglobin Concentration (MCHC) Levels in Blood at Indicated Time Points
Description: Serum MCHC levels were assessed as a clinical hematology laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
g/L
  Day 1; n= 18, 19, 20, 20, 21: number analyzed (Participants) | 18 | 19 | 20 | 20 | 21
  Day 1; n= 18, 19, 20, 20, 21 | 322.9 (13.39) | 321.7 (12.61) | 319.5 (15.36) | 321.5 (12.91) | 327.6 (12.65)
  Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Day 15; n= 17, 19, 17, 21, 21 | 321.5 (11.22) | 324.0 (7.79) | 324.8 (8.35) | 318.3 (12.06) | 322.7 (14.75)
  Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Day 29; n= 16, 19, 17, 18, 17 | 323.3 (14.90) | 329.6 (12.61) | 325.4 (10.25) | 323.6 (8.61) | 323.9 (11.73)
  Day 43; n= 16, 20, 19, 21, 20: number analyzed (Participants) | 16 | 20 | 19 | 21 | 20
  Day 43; n= 16, 20, 19, 21, 20 | 321.9 (13.22) | 325.2 (11.98) | 325.5 (11.23) | 321.0 (11.00) | 327.0 (10.66)

25. Secondary Outcome: Mean Corpuscular Volume (MCV) Levels in Blood at Indicated Time Points
Description: Serum MCV levels were assessed as a clinical hematology laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Femtoliter (fL)
  Day 1; n= 18, 19, 20, 20, 21: number analyzed (Participants) | 18 | 19 | 20 | 20 | 21
  Day 1; n= 18, 19, 20, 20, 21 | 96.7 (5.94) | 96.4 (5.68) | 94.7 (5.28) | 95.7 (4.91) | 96.1 (5.61)
  Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Day 15; n= 17, 19, 17, 21, 21 | 95.9 (6.02) | 95.8 (6.27) | 94.8 (4.53) | 97.0 (6.41) | 98.3 (5.57)
  Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Day 29; n= 16, 19, 17, 18, 17 | 95.8 (5.83) | 95.9 (6.05) | 94.1 (5.94) | 96.3 (4.76) | 97.8 (4.96)
  Day 43; n= 16, 20, 19, 21, 20: number analyzed (Participants) | 16 | 20 | 19 | 21 | 20
  Day 43; n= 16, 20, 19, 21, 20 | 96.1 (5.91) | 95.4 (5.08) | 93.7 (6.09) | 95.6 (5.27) | 97.5 (5.98)

26. Secondary Outcome: Erythrocyte Distribution Width Levels in Blood at Indicated Time Points
Description: Erythrocyte distribution width levels were assessed as a clinical hematology laboratory parameter from Baseline up to follow up visit at Day 43. Day 1 values were considered as Baseline values. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of width
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Percentage of width
  Day 1; n= 18, 19, 20, 20, 21: number analyzed (Participants) | 18 | 19 | 20 | 20 | 21
  Day 1; n= 18, 19, 20, 20, 21 | 15.13 (2.607) | 16.40 (2.082) | 15.41 (1.627) | 15.81 (2.504) | 15.68 (1.725)
  Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Day 15; n= 17, 19, 17, 21, 21 | 15.05 (2.088) | 15.77 (1.569) | 15.26 (1.197) | 16.30 (2.331) | 16.74 (1.912)
  Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Day 29; n= 16, 19, 17, 18, 17 | 15.15 (2.530) | 15.69 (1.750) | 15.36 (1.287) | 15.76 (1.253) | 16.23 (1.668)
  Day 43; n= 16, 20, 19, 21, 20: number analyzed (Participants) | 16 | 20 | 19 | 21 | 20
  Day 43; n= 16, 20, 19, 21, 20 | 15.53 (2.866) | 15.53 (2.018) | 14.95 (1.269) | 15.61 (1.297) | 15.48 (1.389)

27. Secondary Outcome: Change From Baseline in MCH Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including MCH. Change from Baseline in clinical hematology parameters at Day 15, Day 29, Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Pg
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Pg
  Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Day 15; n= 17, 19, 17, 21, 21 | 0.16 (0.602) | 0.19 (0.817) | 0.27 (0.685) | 0.16 (0.520) | 0.25 (0.870)
  Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Day 29; n= 16, 19, 17, 18, 17 | 0.16 (0.982) | 0.58 (1.185) | 0.42 (0.824) | 0.41 (0.744) | 0.15 (0.987)
  Day 43; n= 16, 20, 19, 21, 20: number analyzed (Participants) | 16 | 20 | 19 | 21 | 20
  Day 43; n= 16, 20, 19, 21, 20 | 0.11 (0.981) | 0.13 (0.948) | 0.34 (0.993) | 0.11 (0.842) | 0.29 (0.809)

28. Secondary Outcome: Change From Baseline in MCHC Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including MCHC. Change from Baseline in clinical hematology parameters at Day 15, Day 29, Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
g/L
  Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Day 15; n= 17, 19, 17, 21, 21 | 2.6 (11.09) | 3.0 (14.21) | 3.5 (10.87) | -3.2 (11.48) | -5.0 (12.92)
  Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Day 29; n= 16, 19, 17, 18, 17 | 5.6 (12.81) | 7.3 (16.92) | 7.6 (8.27) | 0.8 (10.04) | -4.4 (12.30)
  Day 43; n= 16, 20, 19, 21, 20: number analyzed (Participants) | 16 | 20 | 19 | 21 | 20
  Day 43; n= 16, 20, 19, 21, 20 | 3.9 (15.92) | 3.0 (16.53) | 6.0 (11.44) | -1.0 (12.12) | -0.3 (9.14)

29. Secondary Outcome: Change From Baseline in MCV Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including MCV. Change from Baseline in clinical hematology parameters at Day 15, Day 29, Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
fL
  Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Day 15; n= 17, 19, 17, 21, 21 | -0.4 (2.98) | -0.2 (3.39) | -0.3 (2.57) | 1.3 (3.15) | 2.2 (3.21)
  Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Day 29; n= 16, 19, 17, 18, 17 | -1.4 (3.24) | -0.5 (2.86) | -0.9 (2.36) | 0.9 (2.54) | 1.6 (2.40)
  Day 43; n= 16, 20, 19, 21, 20: number analyzed (Participants) | 16 | 20 | 19 | 21 | 20
  Day 43; n= 16, 20, 19, 21, 20 | -0.8 (3.15) | -0.7 (3.37) | -0.8 (3.28) | 0.6 (3.06) | 0.9 (2.10)

30. Secondary Outcome: Change From Baseline in Erythrocyte Distribution Width Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including erythrocyte distribution width. Change from Baseline in clinical hematology parameters at Day 15, Day 29, Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Percentage of width
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Percentage of width
  Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Day 15; n= 17, 19, 17, 21, 21 | -0.18 (1.025) | -0.48 (1.276) | -0.09 (1.047) | 0.54 (1.162) | 1.06 (1.337)
  Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Day 29; n= 16, 19, 17, 18, 17 | -0.31 (1.019) | -0.64 (1.332) | -0.23 (1.021) | 0.58 (1.202) | 0.40 (1.342)
  Day 43; n= 16, 20, 19, 21, 20: number analyzed (Participants) | 16 | 20 | 19 | 21 | 20
  Day 43; n= 16, 20, 19, 21, 20 | 0.18 (1.329) | -0.74 (1.728) | -0.50 (1.094) | 0.23 (1.410) | -0.22 (1.165)

31. Secondary Outcome: Change From Baseline in Leukocytes, Neutrophils, Basophils, Eosinophils, Lymphocytes, Monocytes, Platelets Levels
Description: Blood samples were collected from participants to evaluate clinical hematology parameters including leukocytes, neutrophils, basophils, eosinophils, lymphocytes, monocytes, platelets. Change from Baseline in clinical hematology parameters at Day 15, Day 29, Day 43 are presented. Day 1 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
10^12 cells/L
  Leukocytes; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Leukocytes; Day 15; n= 17, 19, 17, 21, 21 | 0.47 (1.271) | -0.21 (1.051) | 0.40 (1.116) | -0.03 (1.476) | -0.03 (1.463)
  Leukocytes; Day 29; n= 16, 19, 17, 18, 17: number analyzed (Participants) | 16 | 19 | 17 | 18 | 17
  Leukocytes; Day 29; n= 16, 19, 17, 18, 17 | 0.49 (1.849) | 0.40 (1.784) | 0.00 (1.084) | -0.14 (1.701) | 0.20 (1.526)
  Leukocytes; Day 43; n= 16, 20, 19, 20, 19: number analyzed (Participants) | 16 | 20 | 19 | 20 | 19
  Leukocytes; Day 43; n= 16, 20, 19, 20, 19 | 0.54 (1.041) | 1.08 (1.662) | 0.23 (1.101) | 0.21 (2.615) | 0.67 (1.580)
  Neutrophils; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Neutrophils; Day 15; n= 17, 19, 17, 21, 21 | 0.391 (1.2323) | -0.146 (0.9163) | 0.280 (1.0681) | 0.259 (1.3874) | 0.344 (1.2469)
  Neutrophils; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Neutrophils; Day 29; n= 16, 18, 17, 17, 15 | 0.237 (1.6283) | 0.469 (1.5717) | -0.021 (1.0157) | -0.009 (1.8718) | 0.273 (1.5729)
  Neutrophils; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Neutrophils; Day 43; n= 16, 20, 19, 19, 19 | 0.423 (1.0535) | 0.904 (1.3737) | 0.112 (1.0449) | 0.504 (2.3110) | 0.691 (1.5221)
  Basophils; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Basophils; Day 15; n= 17, 19, 17, 21, 21 | 0.005 (0.0302) | 0.009 (0.0200) | -0.002 (0.0210) | -0.002 (0.0383) | 0.007 (0.0102)
  Basophils; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Basophils; Day 29; n= 16, 18, 17, 17, 15 | 0.013 (0.0510) | 0.006 (0.0195) | -0.004 (0.0187) | 0.000 (0.0242) | 0.012 (0.0328)
  Basophils; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Basophils; Day 43; n= 16, 20, 19, 19, 19 | 0.006 (0.0268) | 0.001 (0.0148) | -0.004 (0.0203) | -0.001 (0.0228) | 0.007 (0.0192)
  Eosinophils; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Eosinophils; Day 15; n= 17, 19, 17, 21, 21 | 0.009 (0.0698) | -0.017 (0.1313) | -0.006 (0.1345) | -0.006 (0.1183) | -0.053 (0.1478)
  Eosinophils; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Eosinophils; Day 29; n= 16, 18, 17, 17, 15 | 0.020 (0.0859) | -0.002 (0.1226) | -0.006 (0.1129) | 0.025 (0.0990) | 0.007 (0.0880)
  Eosinophils; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Eosinophils; Day 43; n= 16, 20, 19, 19, 19 | 0.061 (0.1193) | 0.030 (0.1439) | 0.051 (0.1647) | 0.021 (0.0984) | -0.024 (0.1876)
  Lymphocytes; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Lymphocytes; Day 15; n= 17, 19, 17, 21, 21 | 0.082 (0.4256) | -0.019 (0.3163) | 0.106 (0.4617) | -0.208 (0.5095) | -0.236 (0.4298)
  Lymphocytes; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Lymphocytes; Day 29; n= 16, 18, 17, 17, 15 | 0.194 (0.6605) | 0.026 (0.4130) | 0.019 (0.4421) | -0.074 (0.7018) | -0.154 (0.3058)
  Lymphocytes; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Lymphocytes; Day 43; n= 16, 20, 19, 19, 19 | 0.018 (0.3427) | 0.061 (0.3332) | 0.007 (0.4824) | -0.064 (0.4759) | -0.041 (0.2801)
  Monocytes; Day 15; n= 17, 19, 17, 21, 21: number analyzed (Participants) | 17 | 19 | 17 | 21 | 21
  Monocytes; Day 15; n= 17, 19, 17, 21, 21 | -0.005 (0.1518) | -0.042 (0.1504) | -0.016 (0.2285) | -0.068 (0.1895) | -0.037 (0.1460)
  Monocytes; Day 29; n= 16, 18, 17, 17, 15: number analyzed (Participants) | 16 | 18 | 17 | 17 | 15
  Monocytes; Day 29; n= 16, 18, 17, 17, 15 | 0.027 (0.1553) | 0.053 (0.1483) | -0.031 (0.2194) | 0.077 (0.2532) | 0.015 (0.1878)
  Monocytes; Day 43; n= 16, 20, 19, 19, 19: number analyzed (Participants) | 16 | 20 | 19 | 19 | 19
  Monocytes; Day 43; n= 16, 20, 19, 19, 19 | 0.033 (0.1631) | 0.065 (0.1629) | 0.026 (0.2652) | -0.021 (0.1855) | 0.023 (0.1249)
  Platelet; Day 15; n= 17, 18, 17, 20, 21: number analyzed (Participants) | 17 | 18 | 17 | 20 | 21
  Platelet; Day 15; n= 17, 18, 17, 20, 21 | -14.2 (26.24) | -16.2 (27.46) | -3.2 (38.13) | -3.3 (27.78) | -10.8 (31.95)
  Platelet; Day 29; n= 16, 18, 17, 17, 17: number analyzed (Participants) | 16 | 18 | 17 | 17 | 17
  Platelet; Day 29; n= 16, 18, 17, 17, 17 | -17.1 (40.58) | -12.8 (36.55) | -18.1 (29.63) | 1.3 (35.58) | -2.4 (33.65)
  Platelet; Day 43; n= 15, 19, 19, 21, 20: number analyzed (Participants) | 15 | 19 | 19 | 21 | 20
  Platelet; Day 43; n= 15, 19, 19, 21, 20 | -4.9 (37.30) | 4.4 (50.34) | -10.4 (35.12) | -1.6 (30.95) | -7.1 (31.95)

32. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings at Indicated Time Points
Description: Single measurements of 12-lead ECG were obtained in supine position using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT interval. Number of participants who had abnormal non clinically significant (NCS) and abnormal clinically significant (CS) ECG findings at Baseline (Week -4) and Day 29 are presented.
Time Frame: Up to Day 29
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Participants
  Baseline(Week -4);Abnormal; NCS;n=19,20,20,22,22 | 10 | 15 | 18 | 12 | 16
  Baseline(Week-4);Abnormal;CS;n=19,20,20,22,22 | 0 | 0 | 0 | 1 | 0
  Day 29; Abnormal; NCS; n=17,19,18,19,17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Day 29; Abnormal; NCS; n=17,19,18,19,17 | 12 | 14 | 16 | 8 | 12
  Day 29; Abnormal; CS; n=17,19,18,19,17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Day 29; Abnormal; CS; n=17,19,18,19,17 | 0 | 0 | 0 | 1 | 0

33. Secondary Outcome: Change From Baseline in ECG Mean Heart Rate
Description: Single measurements of 12-lead ECG were obtained in supine position using an ECG machine to measure HR. Week -4 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values at Day 29 minus Baseline value.
Time Frame: Baseline and Day 29
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
Beats per minute | -2.0 (8.66) | 0.5 (10.53) | 1.1 (7.40) | 2.2 (7.51) | 0.9 (7.09)

34. Secondary Outcome: Change From Baseline in ECG Parameters Including PR Interval, QRS Duration, QT Interval and QTcB
Description: Single measurements of 12-lead ECG were obtained in supine position using an ECG machine to measure PR interval, QRS duration, QT interval and QTcB. Week -4 values were considered as Baseline values. Change from Baseline was calculated by subtracting post-Baseline visit values at Day 29 minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Baseline and Day 29
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Milliseconds (msec)
  PR interval; n= 17, 18, 18, 17, 16: number analyzed (Participants) | 17 | 18 | 18 | 17 | 16
  PR interval; n= 17, 18, 18, 17, 16 | 7.8 (16.86) | 7.3 (12.37) | -3.3 (23.04) | 2.1 (27.13) | -11.5 (24.77)
  QRS duration; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  QRS duration; n= 17, 19, 18, 19, 17 | -1.4 (14.05) | -5.7 (13.36) | -4.7 (47.01) | 1.7 (14.33) | 2.5 (8.97)
  QT interval; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  QT interval; n= 17, 19, 18, 19, 17 | 10.5 (27.16) | 0.7 (31.11) | -19.2 (62.37) | -1.4 (17.72) | -8.2 (33.24)
  QTcB; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  QTcB; n= 17, 19, 18, 19, 17 | 0.0 (30.84) | 5.6 (17.40) | -3.7 (44.86) | 1.1 (20.84) | -5.7 (31.65)

35. Secondary Outcome: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Values at Pre-dialysis and Post-dialysis
Description: Vital sign measurements including SBP and DBP were taken in a seated or semi-supine position in the dialysis chair at specific time points. SBP and DBP were measured pre-dialysis and post-dialysis. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Millimeter of mercury (mmHg)
  SBP; pre-dialysis; Day 1; n= 19, 20, 20, 22, 22 | 142.5 (22.15) | 136.6 (15.39) | 149.2 (26.36) | 144.1 (24.27) | 144.1 (17.01)
  SBP; pre-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  SBP; pre-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 138.8 (24.12) | 138.3 (16.14) | 139.0 (22.77) | 146.6 (20.75) | 142.3 (14.90)
  SBP; pre-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  SBP; pre-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 143.0 (22.08) | 133.1 (18.65) | 143.1 (23.21) | 144.2 (23.27) | 148.7 (19.17)
  SBP; pre-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  SBP; pre-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 140.0 (22.01) | 137.9 (13.21) | 142.0 (24.23) | 149.0 (23.32) | 147.1 (19.18)
  DBP; pre-dialysis; Day 1; n= 19, 20, 20, 22, 22 | 71.9 (14.84) | 68.8 (11.02) | 73.3 (12.96) | 71.8 (14.38) | 72.2 (13.64)
  DBP; pre-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  DBP; pre-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 72.5 (17.76) | 70.0 (11.92) | 70.1 (10.50) | 73.5 (13.69) | 69.7 (12.43)
  DBP; pre-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  DBP; pre-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 70.4 (15.43) | 63.5 (13.55) | 70.9 (12.86) | 73.3 (13.17) | 72.7 (9.96)
  DBP; pre-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  DBP; pre-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 72.5 (14.73) | 66.8 (11.94) | 69.9 (13.54) | 77.9 (16.03) | 72.8 (10.52)
  SBP; post-dialysis; Day 1; n= 19, 20, 20, 22, 22 | 138.6 (18.57) | 137.0 (22.10) | 139.9 (22.24) | 136.7 (21.15) | 140.1 (20.10)
  SBP; post-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  SBP; post-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 138.6 (21.83) | 135.5 (21.63) | 137.7 (23.02) | 137.4 (17.58) | 140.9 (15.34)
  SBP; post-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  SBP; post-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 135.7 (26.04) | 130.1 (18.50) | 133.7 (23.88) | 142.8 (23.96) | 147.8 (19.09)
  SBP; post-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  SBP; post-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 137.5 (22.74) | 135.8 (21.05) | 130.4 (15.47) | 145.2 (20.66) | 137.5 (22.74)
  DBP; post-dialysis; Day 1; n= 19, 20, 20, 22, 22 | 72.1 (15.11) | 67.9 (11.49) | 68.7 (11.64) | 71.1 (12.92) | 71.5 (11.17)
  DBP; post-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  DBP; post-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 72.4 (16.41) | 70.1 (12.84) | 67.8 (11.10) | 71.3 (11.07) | 71.1 (9.51)
  DBP; post-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  DBP; post-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 73.9 (15.11) | 64.4 (9.83) | 67.9 (12.00) | 72.4 (12.43) | 72.9 (11.18)
  DBP; post-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  DBP; post-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 69.5 (15.24) | 67.4 (10.90) | 67.4 (11.24) | 72.9 (12.60) | 75.3 (7.89)

36. Secondary Outcome: Pulse Rate Values at Pre-dialysis and Post-dialysis
Description: Vital sign measurements including pulse rate values were taken in a seated or semi-supine position in the dialysis chair. Pulse rate was measured pre-dialysis and post-dialysis. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Beats per minute
  Pre-dialysis; Day 1; n= 19, 20, 20, 22, 22 | 68.5 (7.95) | 69.9 (9.18) | 66.7 (7.01) | 71.4 (11.25) | 76.5 (9.35)
  Pre-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  Pre-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 76.1 (10.31) | 67.3 (9.20) | 68.3 (7.51) | 72.1 (11.89) | 75.1 (12.68)
  Pre-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Pre-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 70.4 (8.31) | 70.3 (11.54) | 69.6 (9.53) | 70.8 (9.91) | 73.4 (11.45)
  Pre-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  Pre-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 71.5 (9.17) | 69.9 (9.34) | 66.9 (6.74) | 71.3 (10.08) | 75.8 (8.29)
  Post-dialysis; Day 1; n= 19, 20, 20, 22, 22 | 71.0 (11.54) | 68.7 (11.19) | 66.3 (8.37) | 73.2 (12.77) | 78.8 (11.61)
  Post-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  Post-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 72.5 (12.69) | 67.7 (12.24) | 70.1 (12.49) | 73.0 (12.07) | 78.1 (15.72)
  Post-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Post-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 73.6 (7.10) | 69.9 (9.60) | 68.8 (11.29) | 72.2 (9.52) | 77.4 (10.04)
  Post-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  Post-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 72.0 (12.04) | 69.1 (10.21) | 68.0 (10.28) | 71.9 (11.02) | 77.3 (10.26)

37. Secondary Outcome: Weight Values at Post-dialysis
Description: Vital sign measurements including weight values were taken in a seated or semi-supine position in the dialysis chair. Weight was measured post-dialysis. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Kilograms (kg)
  Day 1; n= 19, 20, 20, 22, 22 | 82.38 (25.941) | 80.04 (25.996) | 78.83 (21.331) | 79.38 (23.345) | 76.03 (16.877)
  Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  Day 15; n= 17, 20, 18, 22, 21 | 84.24 (26.652) | 80.00 (25.887) | 79.82 (22.200) | 79.44 (23.500) | 75.55 (17.595)
  Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Day 29; n= 17, 19, 18, 19, 17 | 83.22 (27.198) | 81.04 (25.925) | 80.02 (22.286) | 82.66 (23.036) | 76.07 (18.135)
  Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  Day 43; n= 16, 20, 19, 21, 21 | 83.93 (27.589) | 80.21 (26.683) | 79.25 (21.757) | 80.64 (23.347) | 73.66 (11.614)

38. Secondary Outcome: Change From Baseline in SBP and DBP Values at Pre-dialysis and Post-dialysis
Description: Vital sign measurements including SBP and DBP were taken in a seated or semi-supine position in the dialysis chair. SBP and DBP were measured pre-dialysis and post-dialysis. Pre-dialysis Baseline value was defined as SBP and DBP value obtained pre-dialysis on Day 1. Post-dialysis Baseline value was defined as SBP and DBP value obtained post-dialysis at Week -2. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
mmHg
  SBP; pre-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  SBP; pre-dialysis; Day 15; n= 17, 20, 18, 22, 21 | -2.9 (22.03) | 1.7 (14.14) | -5.6 (14.77) | 2.5 (20.68) | -1.4 (16.35)
  SBP; pre-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  SBP; pre-dialysis; Day 29; n= 17, 19, 18, 19, 17 | -0.6 (20.32) | -3.9 (19.72) | -4.7 (18.17) | 1.3 (17.51) | 4.5 (20.03)
  SBP; pre-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  SBP; pre-dialysis; Day 43; n= 16, 20, 19, 21, 21 | -2.1 (21.34) | 1.2 (17.14) | -6.2 (13.83) | 3.3 (19.47) | 4.3 (10.03)
  SBP; post-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  SBP; post-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 5.4 (21.39) | -3.6 (20.13) | 6.1 (20.81) | 5.7 (21.07) | -0.7 (22.33)
  SBP; post-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  SBP; post-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 2.3 (19.72) | -9.4 (18.50) | 0.8 (24.79) | 9.3 (19.03) | 4.0 (19.76)
  SBP; post-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  SBP; post-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 3.1 (22.22) | -3.2 (21.71) | -3.6 (17.88) | 12.0 (20.19) | 4.7 (20.11)
  DBP; pre-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  DBP; pre-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 1.1 (10.57) | 1.2 (8.85) | -1.7 (9.78) | 1.8 (12.68) | -2.1 (11.04)
  DBP; pre-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  DBP; pre-dialysis; Day 29; n= 17, 19, 18, 19, 17 | -0.3 (11.09) | -4.7 (10.04) | -3.0 (8.99) | 1.4 (10.50) | -0.1 (13.80)
  DBP; pre-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  DBP; pre-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 2.2 (8.80) | -2.0 (9.47) | -3.1 (11.06) | 5.2 (15.08) | 2.1 (11.00)
  DBP; post-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  DBP; post-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 2.4 (11.41) | 2.4 (7.71) | -2.9 (11.11) | 3.6 (9.84) | -0.8 (14.13)
  DBP; post-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  DBP; post-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 3.7 (12.93) | -2.5 (8.52) | -3.2 (11.61) | 4.1 (9.33) | 0.2 (10.59)
  DBP; post-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  DBP; post-dialysis; Day 43; n= 16, 20, 19, 21, 21 | -0.6 (10.07) | -0.3 (9.53) | -3.8 (12.13) | 4.5 (9.99) | 4.8 (10.28)

39. Secondary Outcome: Change From Baseline in Pulse Rate Value at Pre-dialysis and Post-dialysis
Description: Vital sign measurements including pulse rate were taken in a seated or semi-supine position in the dialysis chair. Pulse rate was measured pre-dialysis and post-dialysis. Pre-dialysis Baseline value was defined as pulse rate value obtained pre-dialysis on Day 1. Post-dialysis Baseline value was defined as pulse rate value obtained post-dialysis at Week -2. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
Beats per minute
  Pre-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  Pre-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 7.0 (9.50) | -2.6 (8.46) | 2.3 (5.76) | 0.7 (11.46) | -1.4 (11.15)
  Pre-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Pre-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 2.4 (6.92) | 0.9 (12.86) | 3.4 (7.58) | 0.5 (10.01) | -3.0 (9.14)
  Pre-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  Pre-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 3.1 (9.59) | 0.1 (6.57) | 0.8 (6.11) | -0.6 (10.03) | 0.2 (6.79)
  Post-dialysis; Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  Post-dialysis; Day 15; n= 17, 20, 18, 22, 21 | 2.2 (11.61) | -1.2 (12.86) | 1.1 (10.15) | 0.5 (8.00) | 4.4 (13.28)
  Post-dialysis; Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Post-dialysis; Day 29; n= 17, 19, 18, 19, 17 | 4.2 (9.13) | 1.5 (13.13) | -0.8 (9.79) | 2.6 (9.04) | 6.0 (7.50)
  Post-dialysis; Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  Post-dialysis; Day 43; n= 16, 20, 19, 21, 21 | 2.3 (8.67) | 0.3 (12.96) | -0.8 (9.32) | -0.1 (9.08) | 3.9 (9.32)

40. Secondary Outcome: Change From Baseline in Weight at Post-dialysis
Description: Vital sign measurements including weight were taken in a seated or semi-supine position in the dialysis chair. Weight was measured post-dialysis. Post-dialysis Baseline value was defined as SBP and DBP value obtained post-dialysis at Week -2. Change from Baseline was calculated by subtracting post-Baseline visit values minus Baseline value. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Time Frame: Up to Day 43
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
Number analyzed (Participants) | 19 | 20 | 20 | 22 | 22
kg
  Day 15; n= 17, 20, 18, 22, 21: number analyzed (Participants) | 17 | 20 | 18 | 22 | 21
  Day 15; n= 17, 20, 18, 22, 21 | -0.16 (0.634) | 0.16 (0.971) | -0.01 (0.617) | 0.06 (0.799) | -0.31 (1.215)
  Day 29; n= 17, 19, 18, 19, 17: number analyzed (Participants) | 17 | 19 | 18 | 19 | 17
  Day 29; n= 17, 19, 18, 19, 17 | -0.11 (1.053) | -0.05 (1.583) | -1.23 (5.913) | -0.16 (1.046) | -0.19 (1.244)
  Day 43; n= 16, 20, 19, 21, 21: number analyzed (Participants) | 16 | 20 | 19 | 21 | 21
  Day 43; n= 16, 20, 19, 21, 21 | -0.21 (0.665) | 0.37 (2.760) | -1.39 (5.759) | 0.15 (1.472) | 0.33 (2.169)

ADVERSE EVENTS:
Time Frame: On-therapy serious adverse events (SAEs) and non-serious adverse events (AEs) are presented from the start of study treatment to the end of the 29-day study treatment period plus 1 day, inclusive; an average of 30 days.
Description: On-therapy SAEs and non-serious AEs are reported for members of the safety Population, comprised of all participants who received at least one dose of investigational drug. One participant who was randomized to the placebo group, erroneously received 25mg daprodustat treatment throughout the 29-day treatment period. This subject is counted within the daprodustat 25mg treatment group for all PK population and safety population analyses.
Arm/Group | Placebo | Dapro 10 mg | Dapro 15 mg | Dapro 25 mg | Dapro 30 mg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20 | 0/20 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/19 | 3/20 | 2/20 | 1/22 | 2/22
Other Adverse Events (participants affected / at risk) | 5/19 | 8/20 | 4/20 | 2/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Dapro 10 mg (N=20) | Dapro 15 mg (N=20) | Dapro 25 mg (N=22) | Dapro 30 mg (N=22)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=19) | Dapro 10 mg (N=20) | Dapro 15 mg (N=20) | Dapro 25 mg (N=22) | Dapro 30 mg (N=22)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT02689206/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/06/NCT02689206/SAP_001.pdf